CLINICAL TRIAL: NCT06864988
Title: A Phase 3, Randomized, Double-Masked, Active-Controlled Trial of a Single Intravitreal Injection of 4D-150 in Adults With Macular Neovascularization Secondary to Age-Related Macular Degeneration
Brief Title: 4D-150 in Patients With Macular Neovascularization Secondary to Age-Related Macular Degeneration
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4D-150-C003
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Macular Neovascularization Secondary to Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; AMD; Exudative AMD; Neovascular AMD; Exudative age-related macular degeneration; Neovascular age-related macular degeneration; Wet age-related macular degeneration; Wet macular degeneration; Wet AMD; wAMD; Retinal gene therapy; Intravitreal gene therapy; Genetic Medicine; Ocular Gene Therapy; nAMD
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration | interventions — aflibercept; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4D-150 IVT (3E10 vg/eye) (Experimental)
  Interventions: Biological: 4D-150 IVT (3E10 vg/eye)
- Aflibercept (AFLB) 2 mg IVT (Active Comparator)
  Interventions: Biological: EYLEA® (aflibercept) Injection 2 mg (0.05mL)

INTERVENTIONS:
Biological: 4D-150 IVT (3E10 vg/eye) — If randomized to the 4D-150 treatment arm, 4D-150 will be administered at the assigned dose level as a single dose IVT injection on Day 1
  Arms: 4D-150 IVT (3E10 vg/eye)
Biological: EYLEA® (aflibercept) Injection 2 mg (0.05mL) — Eylea (aflibercept) will be administered at applicable visits
  Arms: Aflibercept (AFLB) 2 mg IVT

SUMMARY:
A Phase 3, Randomized, Double-Masked, Active-Controlled Trial in Adults with Macular Neovascularization Secondary to Age-Related Macular Degeneration

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of age at time of consent
* Treatment naïve MNV secondary to nAMD in the study eye
* Active subfoveal MNV or juxtafoveal/ extrafoveal MNV with a subfoveal component (where activity is defined as evidence of SRF, IRF, subretinal hyperreflective material, or leakage) identified by fluorescein angiography (FA) or spectral domain optical coherence tomography (SD-OCT), in the study eye, at the Screening Visit confirmed by the Reading Center
* Demonstrated clinical response to aflibercept and functional stability in the study eye as confirmed by the Reading Center
* BCVA between 25 and 78 ETDRS letters, inclusive (20/320-20/32 Snellen equivalent) in the study eye at the Screening Visit
* CST less than or equal to 500 microns in the study eye at screening visit, confirmed by the central reading center

Exclusion Criteria:

Ocular Conditions:

* MNV due to causes other than nAMD in either eye (Fibrosis, atrophy, or subretinal hemorrhage in the foveal central subfield (1 mm diameter))
* History of retinal detachment in the study eye
* History of or presence of active inflammation in either eye
* Glaucoma or intraocular hypertension requiring more than 2 topical medications for control

Systemic Conditions and Considerations:

* Major illness or major surgical procedure in the 28 days prior to the Screening Visit
* Uncontrolled blood pressure
* Acute coronary syndrome, myocardial infarction or coronary artery revascularization, cerebrovascular accident, transient ischemic attack within 6 months of the Screening Visit
* History of autoimmune condition that may predispose to the development of uveitis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA ETDRS letter score at Week 52 | 52 Weeks

SECONDARY OUTCOMES:
Mean annualized number of aflibercept injections after Week 4 through Weeks 52 and 104 | 104 Weeks
Incidence and timing of aflibercept injections after Week 4 through Weeks 52 and 104 | 104 Weeks
Proportion of subjects not requiring aflibercept injections after Week 4 through Weeks 52 and 104 in the 4D-150 arm | 104 Weeks
Mean change from baseline in CST over time through Weeks 52 and 104 | 104 Weeks
Mean change from baseline in BCVA ETDRS letter score over time through Weeks 52 and 104 | 104 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hersh Patel, Study Director — 4D Molecular Therapeutics
Locations (101):
- United States (96):
  - Barnet Dulaney Perkins Eye Center, Phoenix, Arizona
  - Retinal Research Institute, LLC, Scottsdale, Arizona
  - Retina Partners of Northwest Arkansas, Springdale, Arkansas
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Retina Associates of Southern California, Huntington Beach, California
  - Loma Linda University Faculty Medical Clinics, Loma Linda, California
  - Jules Stein Eye Institute, Los Angeles, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Gavin Herbert Eye Institute, Orange, California
  - Retina Consultants of San Diego, Poway, California
  - Kaiser Permanente-Riverside Medical Center, Riverside, California
  - Retinal Consultants Medical Group Inc, Sacramento, California
  - Orange County Retina Medical Group, Santa Ana, California
  - California Retina Consultants - Santa Barbara, Santa Barbara, California
  - Bay Area Retina Associates, Walnut Creek, California
  - University of Colorado, Denver, Aurora, Colorado
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - RSC Research, LLC, Denver, Colorado
  - Connecticut Eye Consultants, Danbury, Connecticut
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Vitreo Retinal Associates, Gainesville, Florida
  - Florida Retina Institute - Jacksonville, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Associates of Sarasota, Sarasota, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Georgia Retina PC, Marietta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - University of Chicago, Chicago, Illinois
  - Retina Associates - Elmhurst, Elmhurst, Illinois
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Midwest Eye Institute, Carmel, Indiana
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Haik Humble Eye Center, West Monroe, Louisiana
  - Maine Eye Center, Portland, Maine
  - Wilmer Eye Institute John's Hopkins University, Baltimore, Maryland
  - Retina Group of Washington, Chevy Chase, Maryland
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists - Hagerstown, Hagerstown, Maryland
  - MD Medical Research, Waldorf, Maryland
  - New England Retina Consultants, Springfield, Massachusetts
  - Foundation for Vision Research, Grand Rapids, Michigan
  - Mississippi Retina Associates, Madison, Mississippi
  - Deep Blue Retina Clinical Research, Southaven, Mississippi
  - The Retina Institute, St Louis, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Envision Ocular, LLC, Bloomfield, New Jersey
  - NJ Retina, Edison, New Jersey
  - NJ Retina, Teaneck, New Jersey
  - Eye Associates of New Mexico Vision Research Center, Albuquerque, New Mexico
  - Retina-Vitreous Surgeons of Central New York, Liverpool, New York
  - Vitreous Retina Macula Consultants of New York, New York, New York
  - Retina Associates of Western New York, Rochester, New York
  - Western Carolina Retinal Associate PA, Asheville, North Carolina
  - Duke Eye Center, Durham, North Carolina
  - North Carolina (NC) Retina Associates, Wake Forest, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Piedmont Retina Specialists - Winston Salem Office, Winston-Salem, North Carolina
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Cole Eye Institute, Cleveland, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Verum Research, LLC, Eugene, Oregon
  - EyeHealth Northwest Peterkort, Portland, Oregon
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Erie Retina Research, Erie, Pennsylvania
  - The Scheie Eye Institute, Philadelphia, Pennsylvania
  - Charleston Neuroscience Center, Charleston, South Carolina
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, Knoxville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research, Austin, Texas
  - Retina & Vitreous of Texas, PLLC, Bellaire, Texas
  - Retina Consultants of Houston, Bellaire, Texas
  - Texas Retina Center, Houston, Texas
  - Retina Associates of South Texas PA, San Antonio, Texas
  - Retina Consultants of Texas San Antonio, San Antonio, Texas
  - RCTX - Westover Hills Retina Center, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Strategic Clinical Research Group, LLC, Willow Park, Texas
  - Retina Group of Washington, Fairfax, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia
  - Retina Institute of Virginia, Richmond, Virginia
  - Eye Clinic of Wisconsin, Wausau, Wisconsin
- Canada (5):
  - Calgary Retina Consultants, Calgary, Alberta
  - Retina Surgical Associates, New Westminster, British Columbia
  - St. Michaels Hospital, North York, Ontario
  - Retina Institute of Ottawa, Inc., Ottawa, Ontario
  - Krembil Neuroscience Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided, after deidentification, to qualified researchers with academic interest in AMD in compliance with ICMJE policy. Data or samples shared will be coded, with no Protected Health Information included. Additionally, descriptions of the study protocol, Statistical Analysis Plan (SAP), informed consent and clinical study report may be shared publicly. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party. Data requests can be submitted starting after final Clinical Study Report and the data will be made accessible for a duration determined by the Sponsor, and in accordance with ICMJE policy. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and SAP and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- See also: Related Info — https://4frontclinicalstudies.com